CLINICAL TRIAL: NCT06594302
Title: The Relationship Between Functional Performance and Biopsychosocial Characteristics in Individuals with Systemic Sclerosis
Brief Title: Functional Performance and Biopsychosocial Characteristics in Individuals with Systemic Sclerosis
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Orkun Tüfekçi, Principal Investigator, PT, PhD(c), Hacettepe University
Other Study IDs: SBA 23/171
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Systemic Sclerosis (SSc)
Keywords: functionality; quality of life; biopsychosocial model; BETY-BQ; functional performance; systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Functional performance tests and scales measuring biopsychosocial characteristics — Functional performance tests and scales applications

SUMMARY:
In individuals with systemic sclerosis (SSc), the loss of functionality severely affects quality of life. This condition may cause psychosocial effects by affecting the person, their family, and the environment. Activities of daily living, quality of life, and psychosocial well-being are affected, and aesthetic concerns arise.

Different scales evaluating the quality of life, functions, and disease characteristics of individuals diagnosed with SSc are accepted. In this field, modified Rodnan skin score (mRDS), Duruöz hand index (DHI), scleroderma health assessment questionnaire (SHAQ), and Short Form-36 (SF-36) are frequently used. The BETY-Biopsychosocial Questionnaire is also included in the literature for the evaluation of the biopsychosocial effects of individuals with rheumatism.

In addition, it is essential to evaluate the characteristics of individuals who maintain their health with chronic diseases. Therefore, assessment parameters such as the Chronic Disease Self-Management Scale, Exercise Self-Efficacy Scale, Short Form Illness Perception Scale, Body Awareness Questionnaire, Central Sensitisation Scale, and Tampa Kinesiophobia Questionnaire are frequently used in this regard. The 6 Minute Walk Test (6 MWT) is recommended as a frequently used method to determine cardiopulmonary endurance in individuals with SSc.

It is known that there is a decrease in the distance walked in this test compared to healthy individuals, and the fall potential of physical performance is an important parameter.

In addition, there are also methods used to evaluate physical performance, such as the five-repetition sit-and-stand test (CST), the Stair Climbing Test (SCT), and the Timed up-and-go test (TUG). Considering all these effects, there is a need to examine the relationship between functional and biopsychosocial impact in individuals with SSc.

This study aims to examine the relationship between functional performance and biopsychosocial characteristics in individuals diagnosed with systemic sclerosis and to present the results for this disease group.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Systemic Sclerosis
* To be between 18-65 years old
* Being reader literate

Exclusion Criteria:

* Having a severe musculoskeletal disability
* Being diagnosed with pulmonary hypertension
* History of active infection
* Having a severe neuropsychiatric disorder
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals who come to the university hospital for routine controls.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-10-04 (Estimated)

PRIMARY OUTCOMES:
BETY-Biopsychosocial Questionnaire | Baseline
  The biopsychosocial status of the individual is assessed with questions about pain, functionality, mood, sociability, sexuality, and sleep status. Each question consists of 30 items scored between 0-120 as '0 (never), 1 (yes rarely), 2 (yes sometimes), 3 (yes often), 4 (yes always)'. A high score indicates poor biopsychosocial status
Scleroderma Health Assessment Questionnaire (SHAQ) | Baseline
  It is a scale that evaluates the functionality of individuals diagnosed with systemic sclerosis with a 15 cm long VAS with five complaints about the disease and 20 questions. The total score is scored between 0-3. A high score indicates poor functionality.
6-Minute Walk Test-Borg Scale | Baseline
  To assess the submaximal aerobic capacity of individuals, they will walk for 6 minutes over a distance of 30 meters. The total distance walked in 6 minutes will be recorded in meters. Pulse rate, blood pressure, and oxygen saturation values will be checked before and after the test for the safety of the patients.

SECONDARY OUTCOMES:
Modified Rodnan Skin Score (mRSS) | Baseline
  It is a standard disease activity scoring applied in doctor&amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;#39;s examinations for Systemic Sclerosis patients. It evaluates the skin hardness of 17 different parts of the body. 0= normal skin , 1= mild skin thickness, 2= moderate skin thickness, 3= severe skin thickness. A high score indicates increased skin thickness. The total score is scored between 0-5.
Modified Hand Mobility in Scleroderma (mHAMIS) | Baseline
  It is a method in which a physiotherapist evaluates the hand functions of individuals. Based on observation, it evaluates four different hand functions (finger flexion, finger extension, finger abduction, and dorsal extension of the hand).
Hospital Anxiety and Depression Scale (HADS) | Baseline
  It consists of 14 items, 7 of which assess anxiety, and the other 7 determine depression. Each item is scored between 0 and 3, and the total is scored between 0 and 21. High scores indicate poor anxiety and depression levels.
Duruoz Hand Index | Baseline
  Questionnaire form-18 is a likert-type scale that evaluates different hand functions. It can score between 0-90. A high score means a low hand functions.
Short Form-36 (SF-36) | Baseline
  It is a 36-item, 11-question scale that allows general health screening with eight sub-parameters consisting of general health, physical function, social function, pain, emotional well-being, role limitations due to physical health, role limitations due to emotional problems, and vitality. It is a generic scale; Items are scored as &amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;#39;0 = worst health condition, 100 = best health state&amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;#39;. Each subcategory is scored between 0 and 100 points, with a high score indicating good health.
Chronic Disease Self-Management Scale | Baseline
  The scale, which evaluates the self-management status of the individual with chronic disease, consists of 4 sub-dimensions and 21 items, including Self-Stigmatisation (7 items), Coping with Stigmatisation (5 items), Health Care Effectiveness (5 items) and Treatment Compliance (4 items). The rating of the items in the measurement tool is 1= Never, 2= Rarely, 3= Average, 4= Quite often, and 5= Always.
Exercise Self-Efficacy Scale | Baseline
  The scale consists of 18 items rated from 0% to a maximum power of 100% according to the individual&amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;#39;s self-efficacy for exercise. Participants will record the strength of their efficacy beliefs according to the 100-point scale with 10-unit intervals from 0 (cannot do it) to 50 (moderately able to do it) and 100 (absolutely able to do it).
Brief Illness Perception. Questionnaire | Baseline
  It consists of nine items that express illness perception&amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;#39;s cognitive and emotional representation. In the first eight items, a representation expression related to illness perception is questioned, and each item consists of open-ended answers with a score between 0 and 10. In the last item, the individual is asked to indicate three factors that cause their illness.
Body Awareness Questionnaire | Baseline
  The sensitivity of the individual to normal or abnormal body sensitivity to physical, emotional, and social elements is questioned about sensitivity to physical reactions. The 18-item scale consists of four subgroups (estimation of body reactions, sleep-wake cycle, estimation at the beginning, and attention to changes and responses in the body process). For each of the 18 items, respondents are asked to score between 1 and 7 (1=Not true for me at all, 7=Very true for me). The total score from the questionnaire can be a maximum of 126 and a minimum of 18.
Tampa Scale of Kinesiophobia (TSK) | Baseline
  This consists of 17 statements that assess the subjective rating of kinesiophobia. Statements are rated on a four-point Likert scale from 'strongly disagree' (score 1) to 'strongly agree' (score 4). Four items (4, 8, 11, and 12) are reverse-scored. The total score ranges from 17 to 68, with higher values indicating more severe kinesiophobia.
Central Sensitisation Inventory | Baseline
  It consists of 25 questions evaluating the symptoms associated with central sensitization in 2 parts. Part A of the scale includes questions about symptoms scored between 0-4, and a score above 40 indicates the development of central sensitization. Part B of the scale (no scoring) questions whether the patient has previously received any diagnosis related to one or more central nervous systems.
Five Times Sit to-Stand Test | Baseline
  Assesses lower limb and body strength, power, agility, and ability to get up from a chair and sit down again. The patient sits on a chair with back support and crosses their arms in front of the chest. The patient is asked to stand up and sit down five times as quickly as possible without support from the arms. The time required for five repetitions to sit and stand up is recorded in seconds.
Timed Up and Go Test | Baseline
  The balance status of the individual is evaluated by getting up from a back-supported chair and walking 3 meters at a normal walking speed and returning to the chair and the time of sitting on the chair is measured and recorded in seconds.
Stair Climb Test | Baseline
  To measure the individual^s lower extremity strength and dynamic balance, the time to ascend and descend a 10-step staircase with a handrail in the range of 16-20 cm as fast as possible is recorded in seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Will not be shared to protect the data of individuals